CLINICAL TRIAL: NCT00301210
Title: Assessment of the Level of Physical Dependence and Blockade Efficacy Produced by Tramadol
Brief Title: Assessment of Tramadol as a Treatment for Opioid Addiction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Eric C. Strain, Professor, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-18125-2; R01DA018125-02 (NIH); DPMC
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): tramadol dose 1
  Interventions: Drug: Tramadol
- 2 (Experimental): tramadol dose 2
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Tramadol — oral doses four times per day
  Other Names: Ultram

SUMMARY:
Opioids are one of the most commonly abused drugs among individuals who seek treatment for drug abuse. Thus, it is necessary to develop new treatments for opioid addiction. The purpose of this trial is determine whether tramadol is effective in treating opioid dependent individuals.

DETAILED DESCRIPTION:
This human laboratory study will test the effects of tramadol as a step in its development as a new treatment for opioid dependence. Tramadol is a moderate mu agonist opioid that may produce low levels of opioid physical dependence. Tramadol's capacity for producing physical dependence has not been systematically studied in humans. It is important to quantify tramadol, as it provides a measure of its opioid agonist effects. This would also be informative in regards to the abuse liability of tramadol when used as an analgesic (as currently marketed), or when used in the treatment of opioid addiction (as proposed in this study). The purpose of this trial is to evaluate the level of physical dependence as well as blockade efficacy produced by chronic maintenance on oral tramadol in opioid dependent individuals.

Participants will be randomly assigned to receive different doses of tramadol or placebo for up to six weeks. Experimental sessions will take place up to three times per week during the treatment period. During challenge sessions, participants will receive an injection; four different kinds of effects may occur in a session following this injection. First, no effect may occur (a placebo). Second, an opioid agonist effect may occur (opioid agonists include heroin, morphine, hydromorphone, tramadol, and methadone), which may cause the participant to feel "high." Third, an opioid antagonist effect may occur (e.g., naloxone, naltrexone), which may cause the participant to feel a sense of opioid withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Currently opioid dependent

Exclusion Criteria:

* Significant medical illness (e.g., diabetes mellitus)
* History of seizure
* Current sedative or alcohol dependence
* Pregnant or breastfeeding

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Self-reported effects | up to 4 hours for acute effects
physiologic measures | up to 4 hours for acute effects
observer ratings of effects | up to 4 hours for acute effects
cognitive/performance measures | up to 4 hours for acute effects

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Result] Lanier RK, Lofwall MR, Mintzer MZ, Bigelow GE, Strain EC. Physical dependence potential of daily tramadol dosing in humans. Psychopharmacology (Berl). 2010 Sep;211(4):457-66. doi: 10.1007/s00213-010-1919-3. Epub 2010 Jun 30. PMID 20589494